CLINICAL TRIAL: NCT00003114
Title: Oral Combination Chemotherapy in the Treatment of AIDS-Associated Hodgkin's Disease
Brief Title: Combination Chemotherapy in Treating Patients With AIDS-Related Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU2496; P30CA043703 (NIH); CWRU-2496 (Other: Case Comprehensive Cancer Center); AMC-4A-90; NCI-G97-1351
Record Dates: First submitted 1999-11-01; First posted 2003-08-13 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Lymphoma
Keywords: AIDS-related lymphoma; HIV-associated Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, AIDS-Related | interventions — Filgrastim; Cyclophosphamide; Etoposide; Lomustine; Procarbazine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — Filgrastim (granulocyte colony-stimulating factor) is given subcutaneously on days 5-21 and 33-42.The course is repeated every 6 weeks. A complete or partial response after 1 course of treatment receive two additional courses, but lomustine is omitted in the second course.
Drug: cyclophosphamide — Oral cyclophosphamide on days 22-31. The course is repeated every 6 weeks. A complete or partial response after 1 course of treatment receive two additional courses, but lomustine is omitted in the second course.
Drug: etoposide — Oral etoposide on days 1-3. The course is repeated every 6 weeks. A complete or partial response after 1 course of treatment receive two additional courses, but lomustine is omitted in the second course.
Drug: lomustine — Patients receive oral lomustine on day 1.
Drug: procarbazine hydrochloride — Oral and procarbazine on days 22-31. The course is repeated every 6 weeks. A complete or partial response after 1 course of treatment receive two additional courses, but lomustine is omitted in the second course.
Radiation: radiation therapy — Patients with partial response or stable disease receive radiation therapy and/or continued chemotherapy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with lomustine, etoposide, cyclophosphamide, and procarbazine in treating patients with stage IIB, stage III, or stage IV AIDS-related Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate, response duration, and survival of patients receiving lomustine/etoposide/cyclophosphamide/procarbazine (CECP) for stage IIB-IV AIDS-related Hodgkin's disease.
* Assess the feasibility and toxic effects of CECP in this patient population.

OUTLINE: Patients receive oral lomustine on day 1, oral etoposide on days 1-3, and oral cyclophosphamide and procarbazine on days 22-31. Filgrastim (granulocyte colony-stimulating factor) is given subcutaneously on days 5-21 and 33-42. The course is repeated every 6 weeks.

Patients with a complete or partial response after 1 course of treatment receive two additional courses, but lomustine is omitted in the second course. Patients with partial response or stable disease receive radiation therapy and/or continued chemotherapy. Patients failing to respond after 1 course are removed from the study.

Patients will be followed every 3 months until death.

PROJECTED ACCRUAL: A minimum of 16 evaluable patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IIB-IV AIDS-related Hodgkin's disease

  * Patients with Hodgkin's disease as the only HIV-related condition must have a positive ELISA for HIV confirmed by Western Blot
* Measurable or evaluable disease
* No cytologic or radiologic evidence of CNS involvement

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* ECOG 0-3

Life expectancy:

* At least 6 weeks

Hematopoietic:

* WBC at least 1,500/mm3
* Platelet count at least 50,000/mm3

Hepatic:

* Bilirubin no greater than 3.0 mg/dL

Renal:

* Creatinine no greater than 3.0 mg/dL

Other:

* Active infection is allowed (provided prognosis is estimated to be at least 6 weeks)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for Hodgkin's disease
* At least 4 weeks since chemotherapy for Kaposi's sarcoma

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy for localized stage I or II disease that has progressed beyond initial radiation ports is allowed

Surgery:

* Not specified

Other:

* Concurrent AZT therapy is allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1997-07; Primary Completion 2002-06 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Determine the objective response rate, response duration, and survival of patients receiving lomustine/etoposide/cyclophosphamide/procarbazine (CECP) for stage IIB-IV AIDS-related Hodgkin's disease. | The course is repeated every 6 weeks. Patients will be followed every 3 months until death.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States